CLINICAL TRIAL: NCT02804633
Title: Decreased Opioid Consumption and Enhance Recovery With the Addition of IV-Acetaminophen in Colorectal Patients: A Prospective, Randomized, Double-Blinded, Placebo-Controlled Study
Brief Title: Decrease Opioid Consumption With Intra-Venous (IV) Acetaminophen After Colorectal Surgery (DOCIVA)
Acronym: DOCIVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish Hospital, Cincinnati, Ohio (Other)
Responsible Party: Principal Investigator, Amir H. Aryaie, MD, Jewish Hospital, Cincinnati, Ohio
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: JH 13-04
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Pain Control Post Colorectal Surgery
Keywords: IV acetaminophen; Colorectal Surgery; Enhance Recovery; Opioid Consumption; Pain Management
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IV acetaminophen group (Active Comparator): In addition to PCA (morphine or hydromorphone) all patients receive 1 gram of IV acetaminophen (100 ml ) 30 minutes prior to operation and every 6 hours thereafter for up to 5 days post-operatively or discharge.
  Interventions: Drug: IV Acetaminophen
- Placebo Group (Placebo Comparator): In addition to PCA (morphine or hydromorphone) all patients received placebo (100 ml normal saline) given 30 minutes prior to operation and every 6 hours thereafter for up to 5 days post-operatively or discharge
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IV Acetaminophen — 1 gram every 6 hours
  Arms: IV acetaminophen group
Drug: Placebo — 100 ml of normal saline every 6 hours
  Arms: Placebo Group

SUMMARY:
The investigators hypothesis is that use of IV acetaminophen will significantly decrease use of post-operative opioid consumption and enhances recovery after colorectal surgery.

DETAILED DESCRIPTION:
All patients undergoing laparoscopic and open colorectal surgery are randomized to receive either IV acetaminophen or placebo. All patients received an opioid patient controlled anesthesia (PCA). IV acetaminophen (1 gram) or placebo is given 30 minutes prior to operation and every 6 hours thereafter for up to 5 days post-operatively or discharge.

The investigators primary endpoint is to evaluate opioid consumption during the patient's hospital stay. The investigators secondary endpoints are to evaluate return of gastrointestinal function (ROGIF), time to diet ordered (TTDO), length of hospital stay (LOHS) and occurrence of ileus. Pain is measured with the pain visual analog scale score (PVASS) at 3, 8, 24 and 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing colorectal operation (Hartmann's procedure, sigmoidectomy, left hemicolectomy, right hemicolectomy, transverse colectomy, ileocecectomy, colo-colonic anastomosis, colorectal anastomosis, ileo-colonic anastomosis, low anterior resection, or abdominoperineal resection)
* Age range from 18 to 90 years old
* Patient providing signed, written informed consent before participation in the study

Exclusion Criteria:

* Patient younger than 18 years old or older than 90 years old
* Patient or family is unable to give consent
* Patient who use opioids or tramadol daily for >7 days before study medication administration(patient who, in the investigator's opinion, had or was developing opioid tolerance)
* Patient who had a chronic pain condition or any significant medical disease, laboratory abnormality, or condition that, in the investigator's judgment, could have compromised the subject's welfare, ability to communicate with the study staff, complete study activities, or otherwise restricted study participation
* Patient who had hypersensitivity to opioids, acetaminophen, or the inactive ingredients of the study medication
* Patient who had known or suspected history of alcohol or drug abuse or dependence within the previous 1 year
* Patient who had impaired liver function
* Patient who had fever within first 48 hours post-operatively and required acetaminophen for fever reduction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 48 hours
pain control base on pain visual Analogue Scale Score (1-10) | 48 hours

SECONDARY OUTCOMES:
time to Return of GI function (ROGIF) [Flatus or bowel movement] | through study completion, an average of 5 days
Time to diet ordered (TTDO) | through study completion, an average of 5 days
Length of hospital stay (LOHS) | through study completion, an average of 5 days
Occurrence of ileus | through study completion, an average of 5 days

IPD SHARING:
Plan to Share IPD: Yes